CLINICAL TRIAL: NCT05073458
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Parsaclisib in Participants With Primary Warm Autoimmune Hemolytic Anemia
Brief Title: Study of the Efficacy and Safety of Parsaclisib in Participants With Primary Warm Autoimmune Hemolytic Anemia
Acronym: PATHWAY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A business decision was made to discontinue further enrollment. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 50465-309; 2021-002844-66 (EudraCT Number)
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Warm Autoimmune Hemolytic Anemia (wAIHA)
Keywords: Warm Autoimmune Hemolytic Anemia (wAIHA)
MeSH Terms: interventions — parsaclisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study will be a 24 week double-blind period followed by a 24 week open-label period, followed by a long term extension period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Parsaclisib (Experimental): Participants will receive parsaclisib for 24 weeks (double-blind period). Participant who completed the double-blind period and tolerating the study treatment upon investigator's opinion will continue into open-label period for an additional 24 weeks. Participants may then continue to receive parsaclisib in a long-term extension period.
  Interventions: Drug: parsaclisinib
- Group B: Placebo followed by Parsaclisib (Placebo Comparator): Participants will receive placebo for 24 weeks (double-blind period). Participants who completed the double-blind period will receive parsaclisib in the 24 week open-label period. Participants may then continue to receive parsaclisib in a long-term extension period.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: parsaclisinib — parsaclisib will be administered QD orally
  Other Names: INCB050465
  Arms: Group A: Parsaclisib
Drug: placebo — placebo will be administered QD orally follwed by Parsaclisinib in the open label period
  Arms: Group B: Placebo followed by Parsaclisib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of parsaclisib compared with placebo in participants with Primary Warm Autoimmune Hemolytic Anemia (wAIHA),

DETAILED DESCRIPTION:
Prospective participants must have primary wAIHA as well as other protocol-defined criteria. After participants have been determined to be eligible for the study, they will be randomized to 2:1, with stratification factor of corticosteroid dose and hemoglobin (Hgb <9 g/dL or ≥ 9 g/dL). Once a participant has completed the week 24 assessments in the double-blind period, the participant will have the opportunity to receive parsaclisib in the open-label treatment which will last up to another 24 weeks. Participants may then continue to receive parsaclisib in a long-term extension period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary warm AIHA.
* Participants who have at least 1 unsuccessful prior therapy for warm AIHA or unable to receive or tolerate other therapies.
* Hemoglobin ≥ 6.5 to < 10 g/dL with symptoms of anemia at screening.
* FACIT-F score ≤ 43 at screening.
* Willingness to avoid pregnancy or fathering children.
* Willingness to receive PJP prophylaxis.
* Further inclusion criteria apply.

Exclusion Criteria:

* Women who are pregnant, breastfeeding or who are planning a pregnancy.
* Diagnosis of other types of AIHA (CAD, cold agglutinin syndrome, mixed-type AIHA or paroxysmal cold hemoglobinuria).
* Secondary warm AIHA from any cause or diagnosis of Evans syndrome.
* Splenectomy less than 3 months before randomization.
* Participants with a history or ongoing significant illness as assessed by the investigator.
* Participants with a current of medical history of a malignancy within the past 5 years except basal or squamous cell skin cancer that has been removed and considered cured, or superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy.
* Participants know to be infected with HIV, Hepatitis B, or hepatitis C.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment or exposure to a live vaccine.
* Participants with laboratory values outside of the protocol defined ranges.
* Further exclusion criteria apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (56):
- United States (10):
  - Investigative Site US005, Los Angeles, California
  - Investigative Site US004, Whittier, California
  - Investigative Site US006, Miami, Florida
  - Investigative Site US012, Indianapolis, Indiana
  - Investigative Site US007, The Bronx, New York
  - Investigative Site US002, The Bronx, New York
  - Investigative Site US003, Greenville, North Carolina
  - Investigative Site US009, Canton, Ohio
  - Investigative Site US010, Easton, Pennsylvania
  - Investigative Site US001, Knoxville, Tennessee
- Austria (2):
  - Investigative Site AT002, Salzburg CET
  - Investigative Site AT001, Vienna
- Belgium (2):
  - Investigative Site BE001, La Louvière
  - Investigative Site BE002, Liège
- Investigative Site CA001, Edmonton, Alberta, Canada
- France (3):
  - Investigative Site FR002, Lille
  - Investigative Site FR003, Marseille
  - Investigative Site FR001, Paris
- Germany (2):
  - Investigative Site DE001, Essen
  - Investigative Site DE002, Ulm
- Israel (2):
  - Investigative Site IL002, Haifa
  - Investigative Site IL001, Nahariya
- Italy (6):
  - Investigative Site IT003, Florence
  - Investigative Site IT002, Milan
  - Investigative Site IT001, Novara
  - Investigative Site IT004, Pavia
  - Investigative Site IT006, Rome
  - Investigative Site IT005, Trieste
- Japan (10):
  - Investigative Site JP008, Fukuoka
  - Investigative Site JP004, Isehara
  - Investigative Site JP006, Nagoya
  - Investigative Site JP009, Okayama
  - Investigative Site JP002, Okayama
  - Investigative Site JP010, Osakasayama-shi
  - Investigative Site JP005, Saitama
  - Investigative Site JP007, Sendai
  - Investigative Site JP001, Suita-shi
  - Investigative Site JP003, Tokyo
- Investigative Site NL001, Rotterdam, Netherlands
- Poland (6):
  - Investigative Site PL001, Legnica
  - Investigative Site PL006, Lodz
  - Investigative Site PL003, Nowy Sącz
  - Investigative Site PL005, Opole
  - Investigative Site PL004, Wałbrzych
  - Investigative Site PL002, Wroclaw
- Spain (6):
  - Investigative Site ES006, Badalona
  - Investigative Site ES001, Barcelona
  - Investigative Site ES003, Madrid
  - Investigative Site ES005, Murcia
  - Investigative Site ES004, Tarragona
  - Investigative Site ES002, Valencia
- United Kingdom (5):
  - Investigative Site GB002, Glasgow
  - Investigative Site GB006, London
  - Investigative Site GB003, Norwich
  - Investigative Site GB004, Plymouth
  - Investigative Site GB005, Reading

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was designed to evaluate parsaclisib 2.5 mg QD compared with placebo over a 24-week double-blind treatment period followed by a 24-week open-label treatment period with parsaclisib. Participants could then continue to receive parsaclisib in a long-term extension period.
Groups:
- Parsaclisib: Participants received parsaclisib 2.5 milligrams (mg) once daily (QD) for 24 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period, tolerated study treatment, and, in the investigator's opinion, benefited from treatment had the option of continuing into an open-label treatment period for an additional 24 weeks of parsaclisib 2.5 mg QD, and then the long-term extension period to receive parsaclisib 2.5 mg QD for up to 2 years.
- Placebo Followed by Parsaclisib: Participants received matching placebo QD for 24 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period, tolerated study treatment, and, in the investigator's opinion, benefited from treatment had the option of continuing into an open-label treatment period for 24 weeks of parsaclisib 2.5 mg QD, and then the long-term extension period to receive parsaclisib 2.5 mg QD for up to 2 years. Participants may have received parsaclisib before reaching Week 24.
Period: 24-week Double-blind Period
Arm/Group | Parsaclisib | Placebo Followed by Parsaclisib
Started | 7 | 6
Completed | 4 | 4
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: 24-week Open-label Period
Arm/Group | Parsaclisib | Placebo Followed by Parsaclisib
Started | 4 | 4
Completed | 2 | 2
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 2
Period: Long-term Extension Period (~2 Years)
Arm/Group | Parsaclisib | Placebo Followed by Parsaclisib
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parsaclisib | Placebo Followed by Parsaclisib | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (14.28) | 57.8 (15.54) | 60.23 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 6 | 4 | 10
  Asian | 1 | 1 | 2
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Attaining a Durable Hemoglobin Response
Description: A durable hemoglobin response was defined as hemoglobin ≥10 grams per deciliter (g/dL) with an increase from Baseline of ≥2 g/dL not attributed to rescue therapy at ≥3 of the 4 available visits at Week 12 and/or later during the 24-week double-blind treatment period.
Time Frame: up to Week 24
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug. Treatment groups were determined according to the actual treatment the participant received on Day 1 regardless of assigned study treatment. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received matching placebo QD for 24 weeks during the double-blind treatment period.
Arm/Group | Parsaclisib | Placebo
Number analyzed (Participants) | 3 | 4
percentage of participants | 33.3 | 25.0

2. Secondary Outcome: Percentage of Participants With a ≥3-point Increase From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score at Week 24
Description: The FACIT-F scale was developed to assess anemia-related fatigue. The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days. A clinically meaningful change in the FACIT-F score was defined as ≥3-point increase from Baseline. Item scores range from 0 ("not at all") to 4 ("very much"), and the total score ranges from 0 to 52; lower scores indicate greater fatigue. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib | Placebo
Number analyzed (Participants) | 3 | 4
percentage of participants | 66.7 | 50.0

3. Secondary Outcome: Percentage of Participants With a 50 Meter Increase From Baseline to Week 24 in a 6-minute Walk Test (6MWT)
Description: The 6MWT is used to evaluate submaximal exercise capacity. It is a self-paced measurement of the distance that a participant can quickly walk on a flat, hard surface in a period of 6 minutes.
Time Frame: Baseline; Week 24
Population: Safety Analysis Set. Only participants with available data were analyzed,
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Parsaclisib
Number analyzed (Participants) | 4 | 2
percentage of participants | 0.0 | 100.0

4. Secondary Outcome: Change From Baseline in the FACIT-F Score at Each Post-Baseline Visit
Description: The FACIT-F scale was developed to assess anemia-related fatigue. The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days. A clinically meaningful change in the FACIT-F score was defined as ≥3-point increase from Baseline. Item scores range from 0 ("not at all") to 4 ("very much"), and the total score ranges from 0 to 52; lower scores indicate greater fatigue. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. End of Treatment, Double-blind Period: assessment performed for participants who discontinued treatment before Week 24. End of Treatment, Open-label Period: assessment performed for participants who discontinued treatment after Week 24 and before Week 56. Follow-up Visit 3 occurred 12 weeks after the end of treatment visit.
Time Frame: Baseline; Day 1; Weeks 8, 12, 16, 20, 24, 28, 32, 40, 48, 56, and every 16 weeks post-Week 56
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 6 | 4 | 7
scores on a scale
  Baseline | 28.5 (5.96) | 31.3 (5.12) | 31.1 (7.78)
  Change from Baseline at Week 8: number analyzed (Participants) | 5 | 0 | 5
  Change from Baseline at Week 8 | 8.2 (5.63) |  | 2.4 (7.16)
  Change from Baseline at Week 12: number analyzed (Participants) | 5 | 0 | 5
  Change from Baseline at Week 12 | 7.6 (6.58) |  | 3.6 (8.56)
  Change from Baseline at Week 16: number analyzed (Participants) | 4 | 0 | 5
  Change from Baseline at Week 16 | 3.8 (5.91) |  | 6.2 (7.36)
  Change from Baseline at Week 20: number analyzed (Participants) | 4 | 0 | 2
  Change from Baseline at Week 20 | 2.0 (9.09) |  | 4.5 (7.78)
  Change from Baseline at Week 24: number analyzed (Participants) | 4 | 0 | 3
  Change from Baseline at Week 24 | 3.3 (2.63) |  | 5.0 (5.20)
  Change from Baseline at End of Treatment, Double-blind Period: number analyzed (Participants) | 1 | 0 | 2
  Change from Baseline at End of Treatment, Double-blind Period | 20.0 (NA) — The standard deviation cannot be calculated for a single participant. |  | -8.0 (9.90)
  Change from Baseline at Week 28: number analyzed (Participants) | 0 | 4 | 1
  Change from Baseline at Week 28 |  | 6.5 (6.86) | 6.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 32: number analyzed (Participants) | 0 | 3 | 1
  Change from Baseline at Week 32 |  | -9.0 (13.89) | -1.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 40: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at Week 40 |  | 1.0 (NA) — The standard deviation cannot be calculated for a single participant. |
  Change from Baseline at Week 48: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at Week 48 |  | 5.0 (NA) — The standard deviation cannot be calculated for a single participant. |
  Change from Baseline at End of Treatment, Open-label Period: number analyzed (Participants) | 0 | 1 | 1
  Change from Baseline at End of Treatment, Open-label Period |  | -2.0 (NA) — The standard deviation cannot be calculated for a single participant. | 8.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 56: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at Week 56 |  | 1.0 (NA) — The standard deviation cannot be calculated for a single participant. |
  Change from Baseline at End of Treatment, Long-term Extension Period: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at End of Treatment, Long-term Extension Period |  | 1.0 (NA) — The standard deviation cannot be calculated for a single participant. |
  Change from Baseline at Follow-up Visit 3: number analyzed (Participants) | 0 | 1 | 2
  Change from Baseline at Follow-up Visit 3 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -1.0 (2.83)

5. Secondary Outcome: Percentage Change From Baseline in the FACIT-F Score at Each Post-Baseline Visit
Description: The FACIT-F scale was developed to assess anemia-related fatigue. The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days. A clinically meaningful change in the FACIT-F score was defined as ≥3-point increase from Baseline. Item scores range from 0 ("not at all") to 4 ("very much"), and the total score ranges from 0 to 52; lower scores indicate greater fatigue. Percentage change from Baseline was calculated as ([the post-Baseline value minus the Baseline value]/Baseline value) x 100. End of Treatment, Double-blind Period: assessment performed for participants who discontinued treatment before Week 24. End of Treatment, Open-label Period: assessment performed for participants who discontinued treatment after Week 24 and before Week 56. Follow-up Visit 3 occurred 12 weeks after the end of treatment visit.
Time Frame: Baseline; Day 1; Weeks 8, 12, 16, 20, 24, 28, 32, 40, 48, 56, and every 16 weeks post-Week 56
Population: Safety Analysis Set. Only participants with available data were analyzed,
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 6 | 4 | 7
percentage change
  Week 8: number analyzed (Participants) | 5 | 0 | 5
  Week 8 | 29.6 (21.40) |  | 8.2 (21.25)
  Week 12: number analyzed (Participants) | 5 | 0 | 5
  Week 12 | 28.1 (26.10) |  | 15.30252 (32.05)
  Week 16: number analyzed (Participants) | 4 | 0 | 5
  Week 16 | 12.4 (20.21) |  | 21.9 (27.65)
  Week 20: number analyzed (Participants) | 4 | 0 | 2
  Week 20 | 9.1 (31.07) |  | 12.8 (24.79)
  Week 24: number analyzed (Participants) | 4 | 0 | 3
  Week 24 | 10.1 (6.71) |  | 14.8 (16.97)
  End of Treatment, Double-blind Period: number analyzed (Participants) | 1 | 0 | 2
  End of Treatment, Double-blind Period | 95.2 (NA) — The standard deviation cannot be calculated for a single participant. |  | -32.4 (42.62)
  Week 28: number analyzed (Participants) | 0 | 4 | 1
  Week 28 |  | 22.6 (26.80) | 18.8 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 32: number analyzed (Participants) | 0 | 3 | 1
  Week 32 |  | -26.9 (40.55) | -4.8 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 40: number analyzed (Participants) | 0 | 1 | 0
  Week 40 |  | 2.9 (NA) — The standard deviation cannot be calculated for a single participant. |
  Week 48: number analyzed (Participants) | 0 | 1 | 0
  Week 48 |  | 14.7 (NA) — The standard deviation cannot be calculated for a single participant. |
  End of Treatment, Open-label Period: number analyzed (Participants) | 0 | 1 | 1
  End of Treatment, Open-label Period |  | -5.4 (NA) — The standard deviation cannot be calculated for a single participant. | 25.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 56: number analyzed (Participants) | 0 | 1 | 0
  Week 56 |  | 2.9 (NA) — The standard deviation cannot be calculated for a single participant. |
  End of Treatment, Long-term Extension Period: number analyzed (Participants) | 0 | 1 | 0
  End of Treatment, Long-term Extension Period |  | 2.9 (NA) — The standard deviation cannot be calculated for a single participant. |
  Follow-up Visit 3: number analyzed (Participants) | 0 | 1 | 2
  Follow-up Visit 3 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant | -5.1 (10.41)

6. Secondary Outcome: Change From Baseline in Hemoglobin at Each Post-Baseline Visit
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. End of Treatment, Double-blind Period: assessment performed for participants who discontinued treatment before Week 24. End of Treatment, Open-label Period: assessment performed for participants who discontinued treatment after Week 24 and before Week 56. Follow-up Visits 1, 2, and 3 occurred 4, 8, and 12 weeks, respectively, after the end of treatment visit.
Time Frame: Baseline; Day 1; Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, and every 8 weeks post-Week 56
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 6 | 4 | 7
grams per liter
  Baseline | 86.5 (15.31) | 85.3 (12.97) | 98.4 (21.53)
  Change from Baseline at Week 2: number analyzed (Participants) | 6 | 0 | 7
  Change from Baseline at Week 2 | -9.3 (29.09) |  | 8.7 (11.76)
  Change from Baseline at Week 4: number analyzed (Participants) | 5 | 0 | 6
  Change from Baseline at Week 4 | -4.4 (14.29) |  | 14.2 (13.14)
  Change from Baseline at Week 6: number analyzed (Participants) | 4 | 0 | 7
  Change from Baseline at Week 6 | 2.7 (6.38) |  | 14.3 (16.83)
  Change from Baseline at Week 8: number analyzed (Participants) | 5 | 0 | 5
  Change from Baseline at Week 8 | 12.7 (14.07) |  | 15.0 (18.95)
  Change from Baseline at Week 10: number analyzed (Participants) | 4 | 0 | 6
  Change from Baseline at Week 10 | 16.5 (17.41) |  | 16.5 (16.32)
  Change from Baseline at Week 12: number analyzed (Participants) | 5 | 0 | 6
  Change from Baseline at Week 12 | 13.8 (19.69) |  | 20.5 (11.01)
  Change from Baseline at Week 16: number analyzed (Participants) | 4 | 0 | 5
  Change from Baseline at Week 16 | 19.5 (15.76) |  | 22.4 (16.41)
  Change from Baseline at Week 20: number analyzed (Participants) | 4 | 0 | 3
  Change from Baseline at Week 20 | 15.3 (6.08) |  | 7.7 (1.53)
  Change from Baseline at Week 24: number analyzed (Participants) | 4 | 0 | 3
  Change from Baseline at Week 24 | 19.5 (14.80) |  | 19.3 (22.28)
  Change from Baseline at End of Treatment, Double-blind Period: number analyzed (Participants) | 1 | 0 | 1
  Change from Baseline at End of Treatment, Double-blind Period | -62.4 (NA) — The standard deviation cannot be calculated for a single participant. |  | 11.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 26: number analyzed (Participants) | 0 | 3 | 3
  Change from Baseline at Week 26 |  | 14.0 (9.60) | 3.0 (24.33)
  Change from Baseline at Week 28: number analyzed (Participants) | 0 | 4 | 4
  Change from Baseline at Week 28 |  | 18.9 (19.58) | 8.3 (26.48)
  Change from Baseline at Week 30: number analyzed (Participants) | 0 | 2 | 1
  Change from Baseline at Week 30 |  | 8.1 (32.67) | 27.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 32: number analyzed (Participants) | 0 | 3 | 2
  Change from Baseline at Week 32 |  | 19.0 (31.32) | 26.0 (11.31)
  Change from Baseline at Week 36: number analyzed (Participants) | 0 | 3 | 2
  Change from Baseline at Week 36 |  | 22.8 (18.01) | 18.5 (13.44)
  Change from Baseline at Week 40: number analyzed (Participants) | 0 | 2 | 2
  Change from Baseline at Week 40 |  | 21.5 (12.02) | 26.5 (7.78)
  Change from Baseline at Week 44: number analyzed (Participants) | 0 | 2 | 2
  Change from Baseline at Week 44 |  | 25.0 (21.21) | 27.5 (14.85)
  Change from Baseline at Week 48: number analyzed (Participants) | 0 | 2 | 1
  Change from Baseline at Week 48 |  | 22.5 (21.92) | 32.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at End of Treatment, Open-label Period: number analyzed (Participants) | 0 | 1 | 1
  Change from Baseline at End of Treatment, Open-label Period |  | 127.7 (NA) — The standard deviation cannot be calculated for a single participant. | 124.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 56: number analyzed (Participants) | 0 | 2 | 1
  Change from Baseline at Week 56 |  | 17.5 (12.02) | 36.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at Week 64: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at Week 64 |  | 8.0 (NA) — The standard deviation cannot be calculated for a single participant. |
  Change from Baseline at End of Treatment, Long-term Extension Period: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at End of Treatment, Long-term Extension Period |  | 86.0 |
  Change from Baseline at Follow-up Visit 1: number analyzed (Participants) | 0 | 1 | 4
  Change from Baseline at Follow-up Visit 1 |  | 40.0 (NA) — The standard deviation cannot be calculated for a single participant. | 11.0 (7.62)
  Change from Baseline at Follow-up Visit 2: number analyzed (Participants) | 0 | 1 | 4
  Change from Baseline at Follow-up Visit 2 |  | 32.0 (NA) — The standard deviation cannot be calculated for a single participant. | 12.5 (17.52)
  Change from Baseline at Follow-up Visit 3: number analyzed (Participants) | 0 | 1 | 6
  Change from Baseline at Follow-up Visit 3 |  | 23.0 (NA) — The standard deviation cannot be calculated for a single participant. | 20.3 (9.95)

7. Secondary Outcome: Percentage Change From Baseline in Hemoglobin at Each Post-Baseline Visit
Description: Percentage change from Baseline was calculated as ([the post-Baseline value minus the Baseline value]/Baseline value) x 100. End of Treatment, Double-blind Period: assessment performed for participants who discontinued treatment before Week 24. End of Treatment, Open-label Period: assessment performed for participants who discontinued treatment after Week 24 and before Week 56. Follow-up Visits 1, 2, and 3 occurred 4, 8, and 12 weeks, respectively, after the end of treatment visit.
Time Frame: Baseline; Day 1; Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, and every 8 weeks post-Week 56
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 6 | 4 | 7
percentage change
  Week 2: number analyzed (Participants) | 6 | 0 | 7
  Week 2 | -12.3 (41.18) |  | 8.2 (13.82)
  Week 4: number analyzed (Participants) | 5 | 0 | 6
  Week 4 | -3.5 (16.87) |  | 14.2 (13.68)
  Week 6: number analyzed (Participants) | 4 | 0 | 7
  Week 6 | 3.4 (7.42) |  | 14.2 (18.21)
  Week 8: number analyzed (Participants) | 5 | 0 | 5
  Week 8 | 14.0 (14.59) |  | 14.3 (19.65)
  Week 10: number analyzed (Participants) | 4 | 0 | 6
  Week 10 | 17.8 (17.44) |  | 16.5 (17.59)
  Week 12: number analyzed (Participants) | 5 | 0 | 6
  Week 12 | 13.6 (21.15) |  | 20.7 (12.36)
  Week 16: number analyzed (Participants) | 4 | 0 | 5
  Week 16 | 21.7 (16.02) |  | 23.2 (17.81)
  Week 20: number analyzed (Participants) | 4 | 0 | 3
  Week 20 | 18.5 (9.32) |  | 7.6 (2.11)
  Week 24: number analyzed (Participants) | 4 | 0 | 3
  Week 24 | 22.7 (15.52) |  | 19.4 (22.70)
  Change from Baseline at End of Treatment, Double-blind Period: number analyzed (Participants) | 1 | 0 | 1
  Change from Baseline at End of Treatment, Double-blind Period | -87.9 (NA) — The standard deviation cannot be calculated for a single participant. |  | 12.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 26: number analyzed (Participants) | 0 | 3 | 3
  Week 26 |  | 15.2 (9.34) | 3.4 (24.52)
  Week 28: number analyzed (Participants) | 0 | 4 | 4
  Week 28 |  | 23.4 (25.16) | 9.7 (27.56)
  Week 30: number analyzed (Participants) | 0 | 2 | 1
  Week 30 |  | 6.6 (36.17) | 30.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 32: number analyzed (Participants) | 0 | 3 | 2
  Week 32 |  | 23.6 (40.57) | 29.0 (12.41)
  Week 36: number analyzed (Participants) | 0 | 3 | 2
  Week 36 |  | 29.3 (26.69) | 20.6 (14.85)
  Week 40: number analyzed (Participants) | 0 | 2 | 2
  Week 40 |  | 29.7 (18.67) | 29.6 (8.46)
  Week 44: number analyzed (Participants) | 0 | 2 | 2
  Week 44 |  | 34.9 (31.46) | 30.7 (16.35)
  Week 48: number analyzed (Participants) | 0 | 2 | 1
  Week 48 |  | 31.6 (32.12) | 35.6 (NA) — The standard deviation cannot be calculated for a single participant.
  Change from Baseline at End of Treatment, Open-label Period: number analyzed (Participants) | 0 | 1 | 1
  Change from Baseline at End of Treatment, Open-label Period |  | 31.7 (NA) — The standard deviation cannot be calculated for a single participant. | 25.3 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 56: number analyzed (Participants) | 0 | 2 | 1
  Week 56 |  | 24.3 (18.21) | 40.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Week 64: number analyzed (Participants) | 0 | 1 | 0
  Week 64 |  | 10.1 (NA) — The standard deviation cannot be calculated for a single participant. |
  Change from Baseline at End of Treatment, Long-term Extension Period: number analyzed (Participants) | 0 | 1 | 0
  Change from Baseline at End of Treatment, Long-term Extension Period |  | 8.9 (NA) — The standard deviation cannot be calculated for a single participant. |
  Follow-up Visit 1: number analyzed (Participants) | 0 | 1 | 4
  Follow-up Visit 1 |  | 41.2 (NA) — The standard deviation cannot be calculated for a single participant. | 11.5 (8.19)
  Follow-up Visit 2: number analyzed (Participants) | 0 | 1 | 4
  Follow-up Visit 2 |  | 33.0 (NA) — The standard deviation cannot be calculated for a single participant. | 14.5 (19.47)
  Follow-up Visit 3: number analyzed (Participants) | 0 | 1 | 6
  Follow-up Visit 3 |  | 23.7 (NA) — The standard deviation cannot be calculated for a single participant. | 23.4 (13.52)

8. Secondary Outcome: Percentage of Participants Who Received Transfusions From Week 6 to Week 24 and From Week 24 to Week 48
Description: Transfusion was permitted as a rescue treatment. Rescue medication was to be considered if the absolute hemoglobin level continued to decline, there was a > 1 g/dL decrease in hemoglobin from the prior assessment, or the participant developed new or worsening symptoms of warm autoimmune hemolytic anemia (wAIHA).
Time Frame: Week 6 to Week 24; Week 24 to Week 48
Population: Safety Analysis Set. Only participants with available data were analyzed. The number of participants analyzed at Weeks 6 to 24 reflects the number of participants who received study drug for at least 43 days. The number of participants analyzed at Weeks 24 to 48 reflects the number of participants who received study drug during the open-label period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 5 | 4 | 7
percentage of participants
  Week 6 to Week 24: number analyzed (Participants) | 5 | 0 | 7
  Week 6 to Week 24 | 0.0 |  | 42.9
  Week 24 to Week 48: number analyzed (Participants) | 0 | 4 | 4
  Week 24 to Week 48 |  | 25.0 | 25.0

9. Secondary Outcome: Change From Baseline in Daily Corticosteroid Dose at Week 24
Description: A new or increased dose of corticosteroids (prednisone or equivalent) from the Day 1 dose was permitted as rescue treatment. Rescue medication was to be considered if the absolute hemoglobin level continued to decline, there was a > 1 g/dL decrease in hemoglobin from the prior assessment, or the participant developed new or worsening symptoms of wAIHA. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo | Parsaclisib
Number analyzed (Participants) | 3 | 6
milligrams
  Baseline | 13.3 (5.77) | 20.8 (10.21)
  Change from Baseline at Week 24: number analyzed (Participants) | 3 | 5
  Change from Baseline at Week 24 | 8.1 (14.02) | -4.8 (10.41)

10. Secondary Outcome: Percentage Change From Baseline in Daily Corticosteroid Dose at Week 24
Description: A new or increased dose of corticosteroids (prednisone or equivalent) from the Day 1 dose was permitted as rescue treatment. Rescue medication was to be considered if the absolute hemoglobin level continued to decline, there was a > 1 g/dL decrease in hemoglobin from the prior assessment, or the participant developed new or worsening symptoms of wAIHA. Percentage change from Baseline was calculated as ([the post-Baseline value minus the Baseline value]/Baseline value) x 100.
Time Frame: Baseline; Week 24
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Parsaclisib
Number analyzed (Participants) | 3 | 5
percentage change | 81.0 (140.21) | -22.0 (60.07)

11. Secondary Outcome: Percentage of Participants Who Required Rescue Therapy at Any Visit From Week 6 Through Week 24, and From Week 24 to Week 48
Description: Rescue medication was to be considered if the absolute hemoglobin level continued to decline, there was a > 1 g/dL decrease in hemoglobin from the prior assessment, or the participant developed new or worsening symptoms of wAIHA.
Time Frame: Week 6 to Week 24; Week 24 to Week 48
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 5 | 4 | 7
percentage of participants
  Week 6 to Week 24: number analyzed (Participants) | 5 | 0 | 7
  Week 6 to Week 24 | 0.0 |  | 0.0
  Week 24 to Week 48: number analyzed (Participants) | 0 | 4 | 4
  Week 24 to Week 48 |  | 0.0 | 20.0

12. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. An AE could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. TEAEs were defined as AEs reported for the first time or the worsening of pre-existing events after the first dose of study drug.
Time Frame: up to 446 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 6 | 4 | 7
Participants | 4 | 4 | 7

13. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. TEAEs were defined as AEs reported for the first time or the worsening of pre-existing events after the first dose of study drug. The severity of AEs were assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 446 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Placebo Followed by Parsaclisib | Parsaclisib
Number analyzed (Participants) | 6 | 4 | 7
Participants | 1 | 3 | 6

ADVERSE EVENTS:
Time Frame: up to 446 days
Description: For safety analysis, participants who transitioned from treatment with placebo to treatment with parsaclisib 2.5 milligrams (mg) once daily (QD) in the the open-label treatment period and the long-term extension period have been counted both in the placebo arm and the parsaclisib arm.
Groups:
- Placebo: Participants received matching placebo QD for 24 weeks during the double-blind treatment period. Participants who completed the double-blind treatment period, tolerated study treatment, and, in the investigator's opinion, benefited from treatment had the option of continuing into an open-label treatment period for 24 weeks of parsaclisib 2.5 mg QD, and then the long-term extension period to receive parsaclisib 2.5 mg QD for up to 2 years. Participants may have received parsaclisib before reaching Week 24.
Arm/Group | Placebo | Parsaclisib
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/6 | 6/11
Other Adverse Events (participants affected / at risk) | 4/6 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Parsaclisib (N=11)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Parsaclisib (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choluria (Renal and urinary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT05073458/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05073458/SAP_001.pdf